CLINICAL TRIAL: NCT03811808
Title: Multiple System Atrophy Multidisciplinary Clinic
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Steven Vernino MD PhD, PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU 082015-008
Record Dates: First submitted 2017-12-05; First posted 2019-01-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Multiple System Atrophy (MSA)
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MSA patients: patients diagnosed with possible or probable multiple system atrophy

SUMMARY:
This is a prospective cohort study to examine the disease burden of multiple system atrophy and the impact of multidisciplinary care on quality of life and caregiver burden. Data will be collected through valid rating scales completed by patients and caregivers at home or in the MSA clinic.

DETAILED DESCRIPTION:
Study Procedures:

Participants and caregivers will attend a multidisciplinary MSA clinic one day every four months. In addition to the standard of care, they will be asked to complete both online and paper questionnaires, including the following:

* UMSARS (Unified MSA Rating Scale)
* MSA QOL
* CES-D
* OHQ
* Compass-31
* BIC
* UPDRS
* SARA
* MDS Scale
* CGI
* MoCA

Participants will be part of the study as long as they are a patient of the MSA clinic, and will be contacted for follow-up information up to five years.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a patient in the UT Southwestern MSA clinic and be able to attend the multidisciplinary clinic every 4 months
* Patients with possible or probable MSA based on established criteria
* Subjects must be 18 years or older

Exclusion Criteria:

* Patients that are unable to give consent
* Minor patients (younger than age 18)
* Non-English speaking patients
* Subjects that are diagnosed with dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years or older with diagnosis of possible or probable MSA
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Multiple System Atrophy-Quality of Life (MSA-QoL) | at 5 year evaluation
  The disease burden of MSA and impact of multidisciplinary care on the quality of life of patients as measured by the MSA-Quality of Life (QOL) questionnaire completed every four months by the patients. The scale measures how MSA affects a person's quality of life in day to day activities. The scale ranges from No problem to Extreme Problem. The More Extreme Problem sections selected the more their quality of life is affected by the disease.

SECONDARY OUTCOMES:
Unified Multiple System Atrophy Rating Scale (UMSARS) | at 5 year evaluation
  The UMSARS completed every four months by the physician. The scale measures how MSA has progressed from baseline. The higher the score the higher the progression is.
Caregiver Burden Index/ The Zarit Burden Interview | at 5 year evaluation
  The disease burden of MSA and impact of multidisciplinary care on caregiver burden as measured by the Burden Index of Caregivers (BIC) questionnaire and The Zarit Burden Interview completed every four months by the caregivers. The higher the higher the score the more burden the caregiver has.

OTHER OUTCOMES:
Composite Autonomic Symptom Score (CONPASS 31) | at 5 year evaluation
  Compass 31 scale includes 31 questions and it will be used to assess autonomic symptoms that provides clinically relevant scores of autonomic symptom severity based. The higher the score the more autonomic symptoms present
Center for Epidemiologic Studies Depression Scale (CES-D) | at 5 year evaluation
  The CES-D measures symptoms defined by the American Psychiatric Association' Diagnostic and Statistical Manual (DSM-V) for a major depressive episode. The higher the scores and indicative for depression present.
The Orthostatic Hypotension Questionnaire (OHQ) | at 5 year evaluation
  The OHQ is used to assess the comprehensive symptom burden and severity of neurogenic orthostatic hypotension (NOH).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Vernino, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No